CLINICAL TRIAL: NCT04018365
Title: A Multicenter, Open-label, Single-arm Study With Regard to the Efficacy and Safety of Empagliflozin in Patients With Refractory Diabetes Mellitus With Insulin Resistance
Brief Title: A Study of Empagliflozin in Patients With Refractory Diabetes Mellitus With Insulin Resistance
Acronym: EMPIRE-01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kobe University (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Wataru Ogawa, Professor, Division of Diabetes and Endocrinology, Kobe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190012
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Insulin Resistance - Type A; Insulin Resistance - Type B; Lipoatrophic Diabetes Mellitus; Insulin Resistance Syndrome
Keywords: insulin resistance; refractory diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Resistant, with Acanthosis Nigricans; Diabetes Mellitus, Lipoatrophic; Metabolic Syndrome; Insulin Resistance; Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment of empagliflozin (Experimental): Empagliflozin 10 mg is to be continuously administered once daily for 12 weeks. Measure an HbA1c level after 12 weeks and determine the dose (Week 13 to Week 24). In case of <7.0%, 10 mg will be continued: in case of >=7.0%, it will be increased to 25 mg.
  Interventions: Drug: Empagliflozin Tablets

INTERVENTIONS:
Drug: Empagliflozin Tablets — The administration is oral administration with water before or after breakfast.
  Other Names: BI10773

SUMMARY:
A multicenter, open-label, single-arm study with regard to the efficacy and safety of empagliflozin in patients with refractory diabetes mellitus with insulin resistance

DETAILED DESCRIPTION:
To evaluate the clinical efficacy of a treatment with empagliflozin in refractory diabetes mellitus patients with insulin resistance (insulin resistance syndrome, lipoatrophic diabetes mellitus) by using the HbA1c change at Week 24 of treatment from baseline

ELIGIBILITY:
Inclusion Criteria:

* 1) A patient who has been diagnosed with insulin resistance syndrome (type A, type B, type non-A non-B) or lipoatrophic diabetes mellitus prior to obtaining consent
* 2) A patient who has received consistent dosage and administration of drugs aiming a hypoglycemic effect and consistent instructions of diet therapy/exercise therapy for more than 12 weeks before enrollment
* 3) A patient with >= 7.0 % of HbA1c at the time of screening
* 4) A patient, if taking other SGLT2 inhibitor than empagliflozin, whose SGLT2 inhibitor can be washed out for more than 12 weeks prior to starting empagliflozin
* 5) A patient at the age of >=20 years at the time of consent
* 6) A patient who has received sufficient explanation with regard to information such as the objectives and details of this study, expected drug efficacy/pharmacological action, and risks, and has given written consent by her/himself.

Exclusion Criteria:

* 1) A patient with a medical history of acute coronary syndrome (including non-ST-elevation myocardial infarction, ST-elevation myocardial infarction, and unstable angina pectoris), stroke or transient ischemic attack (TIA) within 3 months before obtaining consent
* 2) A patient with suspected hepatic dysfunction, that either of serum ALT, AST or alkaline phosphatase in the screening period is exceeding 3-fold of upper limit of normal rang
* 3) A patient who is receiving a systemic steroid at the time of consent (except for type B)
* 4) A patient whose thyroid hormone product dose has been changed within 6 weeks before obtaining consent
* 5) A patient with unstable endocrine diseases other than diabetes mellitus
* 6) A patient with hemolysis or blood diseases that destabilize erythrocytic cells and other various disorders (e.g., malaria, babesiosis, hemolytic anemia).
* 7) A premenopausal female patient (the latest menstruation was within 1 year before obtaining consent), a lactating or pregnant patient, or a patient who may be pregnant (without hysterectomy or ovariectomy) who has no intention to use efficacious contraception defined in this study during the treatment period and would not agree to receive regular pregnancy tests during the treatment period
* 8) A patient who has experienced alcohol abuse or drug abuse within 3 months before obtaining consent, which may disturb the study participation
* 9) A patient who is in the condition that makes it difficult to administer the study drug
* 10) A patient with renal dysfunction of eGFR (MDRD calculating formula) < 45 mL/min/1.73 m2 in the screening period
* 11) A patient who indicates a hypersensitivity response to empagliflozin or its excipients, or a patient with lactose-intolerance
* 12) A patient with severe ketosis, diabetic coma or precoma, severe infection, perioperative status, or serious trauma
* 13) A patient that the investigator and/or subinvestigator, etc., has judged to be ineligible to this study for other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c change at Week 24 of the treatment from baseline | at Week 24 of the treatment from baseline
  With regard to the HbA1c change at Week 24 of the treatment from baseline, changes will be shown by patient, as well as summarizing with the size of sample, mean, standard deviation, minimum, median, and maximum.

SECONDARY OUTCOMES:
HbA1c change rate at Week 24 of the treatment from baseline | at Week 24 of the treatment from baseline
  With regard to the HbA1c change rate at Week 24 of the treatment from baseline, change rates will be shown by patient, as well as summarizing with the size of sample, mean, standard deviation, minimum, median, and maximum.
HbA1c change at Week 12 of the treatment from baseline | at Week 12 of the treatment from baseline
  With regard to the HbA1c change at Week 12 of the treatment from baseline, changes will be shown by patient, as well as summarizing with the size of sample, mean, standard deviation, minimum, median, and maximum.
HbA1c over time | at Week 24 of the treatment from baseline
  The HbA1c level at measurement time point is tabulated by patient, as well as plotting the HbA1c level over time by line graph. In addition, the mean, standard deviation, interquartile range, minimum, median, and maximum of HbA1c at each time point will be calculated and tabulated, as well as displaying the mean at each measurement time point with error bar of standard deviation by line graph.
Fasting plasma glucose (FPG) over time | at Week 24 of the treatment from baseline
  The FPG level at measurement time point is tabulated by patient, as well as plotting the FPG level over time by line graph. In addition, the mean, standard deviation, interquartile range, minimum, median, and maximum of FPG at each time point will be calculated and tabulated, as well as displaying the mean at each measurement time point with error bar of standard deviation by line graph.
FPG change at Week 24 of the treatment from baseline | at Week 24 of the treatment from baseline
  With regard to the FPG change at Week 24 of the treatment from baseline, changes will be shown by patient, as well as summarizing with the size of sample, mean, standard deviation, minimum, median, and maximum.
Change of insulin dose | at Week 24 of the treatment from baseline
  The insulin dose of each patient will be tabulated by time point.
Postprandial glucose for 2 hours over time | 2 Weeks from Day0 and Day140
  The postprandial glucose for 2 hours at measurement time point is tabulated by patient, and the glucose level over time is plotted by line graph. In addition, the mean, standard deviation, interquartile range, minimum, median, and maximum of postprandial glucose for 2 hours at each time point will be tabulated, and the mean at each measurement time point with an error bar of standard deviation will be displayed by line graph.

CONTACTS AND LOCATIONS:
Overall Officials: Wataru Ogawa, Study Chair — Kobe University Hospital
Locations (5):
- Japan (5):
  - Kobe University Hospital, Kobe, Hyōgo
  - Tohoku University Hospital, Sendai, Miyagi
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - NIhon University Hospital, Chiyoda-ku, Tokyo
  - Okayama University Hospital, Okayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirota Y, Kakei Y, Imai J, Katagiri H, Ebihara K, Wada J, Suzuki J, Urakami T, Omori T, Ogawa W. A Multicenter, Open-Label, Single-Arm Trial of the Efficacy and Safety of Empagliflozin Treatment for Refractory Diabetes Mellitus with Insulin Resistance (EMPIRE-01). Diabetes Ther. 2024 Feb;15(2):533-545. doi: 10.1007/s13300-023-01526-x. Epub 2024 Jan 13. PMID 38216831